CLINICAL TRIAL: NCT03238937
Title: Treatment of Central Sleep Apnea in Patients With Heart Failure With a Cervically Implanted Phrenic Nerve Stimulator
Brief Title: Phrenic Nerve Stimulation for Treatment of Central Sleep Apnea
Acronym: STIMULATE-CSA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No eligible subjects were identified.
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Responsible Party: Principal Investigator, Lana Tsao, Cardiologist, Steward St. Elizabeth's Medical Center of Boston, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00745
Record Dates: First submitted 2017-07-17; First posted 2017-08-03 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Sleep Apnea, Central; Heart Failure
MeSH Terms: conditions — Sleep Apnea, Central; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Phrenic Nerve Stimulator (Other): Phrenic Nerve Stimlator
  Interventions: Device: Phrenic nerve stimulator
- no intervention (No Intervention): Patients without phrenic nerve stimulation

INTERVENTIONS:
Device: Phrenic nerve stimulator — Implantation of phrenic nerve stimulator
  Other Names: no intervention / medical management only
  Arms: Phrenic Nerve Stimulator

SUMMARY:
The study objectives are to demonstrate the ease and safety of bilateral cervically implanted phrenic nerve stimulators for Central Sleep Apnea in patients with Heart Failure. To demonstrate the efficacy, both in the short and long term, of implanted phrenic nerve stimulators in patients with Central Sleep Apnea and Heart Failure. Central Sleep Apnea is a form of hypoventilation syndrome, for which this device is FDA approved. We will also determine if the patient's quality and duration of life is improved by using the PNS to treat CSA in heart failure patients.

DETAILED DESCRIPTION:
This is a multi-center prospective cohort study to monitor the effect of bilateral phrenic nerve stimulation for treatment of central sleep apnea (CSA) in patients with heart failure. There will be 2 groups of study patients, both with CSA and heart failure. One group will receive the phrenic nerve pacer, and one will not. Both groups will have the same medical oversight, management, and assessment of heart health whether they receive the pacer or not.

Subjects will have a physical exam, review of medications, New York Heart Association (NYHA) functional classification assessment for heart failure, Minnesota Living With Heart Failure (MLWHF) Questionnaire for quality of live assessment and blood test for Pro-BNP. In-lab sleep study will be required if subject haven't had one within 3 months, and Echocardiogram, if subjects haven't had one within 30 days. If subjects are willing to have stimulator placement procedure, they'll have an ENT consult. Subjects in the procedure arm will have Phrenic Nerve Stimulator placement procedure, and 3 weeks after procedure follow up visit with ENT doctor to activate the device and have sleep study to confirm proper settings.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female, age 18 to 80 years inclusive.

  2. New York Heart Association (NYHA) class III or IV, or NYHA class II with an episode of heart failure requiring hospitalization in the past 24 months.

  3. Stable on guide line directed medical therapy (GDMT) for 30 days prior to enrollment.

  4. Moderate or severe sleep apnea, that is an Apnea Hypopnea Index (AHI) of >15/hour with >50% being central apneas.

  5. Willing and able to provide written informed consent in compliance with the regulatory requirements. If a subject is unable to provide written informed consent, written informed consent may be obtained from the subject's legal representative.

Exclusion Criteria:

1. Phrenic nerve palsy.
2. Baseline hypoxia (oxygen saturation <90% on room air).
3. On supplemental oxygen.
4. Severe COPD.
5. Unstable angina, MI or cardiac procedure within 3 months of phrenic nerve stimulator placement.
6. Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the protocol.
7. Any other reasons that, in the opinion of the Investigator, the candidate is determined to be unsuitable for entry into the study.

   -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment related adverse events as assessed by CTCAEv40 | 2 years
  Visual Analog Score for pain, BMI in Kg/m ^2

SECONDARY OUTCOMES:
Improvement in quality of life with phrenic nerve stimulation in patients with central sleep apnea and heart failure | 2 years
  Physicians Global Assessments to measure quality of life,

CONTACTS AND LOCATIONS:
Overall Officials: Lana Tsao, MD, Principal Investigator — Steward St. Elizabeth's Medical Center
Locations (1):
- SEMC, Brighton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share protocol and study results
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: once the protocol is approved and as data becomes available indefinitively
Access Criteria: via secure website